CLINICAL TRIAL: NCT01913535
Title: Double-Blind, Placebo-Controlled, Proof-of-Concept (POC) Trial of CERC-501, a Kappa-Selective Opioid Receptor Antagonist, Augmentation of Antidepressant Therapy in Treatment-Resistant Depression (TRD)
Brief Title: Proof-of-Concept Trial of CERC-501 Augmentation of Antidepressant Therapy in Treatment-Resistant Depression
Acronym: RAPID KOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Butler Hospital (Other); Rush University (Other); Temple University (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Overall Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP-002; 271201100006I-0-27100007-1 (NIH)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; Treatment Resistant Depression; Antidepressant; Major Depression; MDD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Depressive Disorder, Major | interventions — Aticaprant

STUDY DESIGN:
Intervention Model Description: sequential parallel comparison design (SPCD) with two phases
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Low Dose Drug-Drug Arm (Active Comparator): Patients in this arm will receive CERC-501 10.0 mg/day for 3 days (in Phase 1) and for 3 subsequent days (in Phase 2)
  Interventions: Drug: CERC-501
- High Dose Drug-Drug Arm (Active Comparator): Patients in this arm will receive CERC-501 20.0 mg/day for 3 days (in Phase 1) and for 3 subsequent days (in Phase 2)
  Interventions: Drug: CERC-501
- Placebo/Low-Dose Drug Arm (Other): Patients in this arm will receive placebo for 3 days (in Phase 1) and CERC-501 10.0 mg/day for 3 days (in Phase 2)
  Interventions: Drug: CERC-501; Drug: Placebo
- Placebo/High-Dose Drug Arm (Other): Patients in this arm will receive placebo for 3 days (in Phase 1) and CERC-501 20.0 mg/day for 3 days (in Phase 2)
  Interventions: Drug: CERC-501; Drug: Placebo
- Placebo/Placebo Arm (Placebo Comparator): Patients in this arm will receive placebo for 3 days (in Phase 1) and for 3 subsequent days (in Phase 2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CERC-501 — Low dose of CERC-501 will be 10 mg/day during the first phase (3 days) and during the second phase (3 days).
  High Dose of CERC-501 will be 20 mg/day during the first phase (3 days) and during the second phase (3 days).
  For patients randomly assigned to the placebo/low-dose drug sequence, the patient will receive placebo for 3 days and then 10 mg/day CERC-501 for the following 3 days.
  For patients randomly assigned to the placebo/high-dose drug sequence, the patient will receive placebo for 3 days and then 20 mg/day CERC-501 for the following 3 days.
  Arms: High Dose Drug-Drug Arm; Low Dose Drug-Drug Arm; Placebo/High-Dose Drug Arm; Placebo/Low-Dose Drug Arm
Drug: Placebo — For patients randomly assigned to the placebo/ placebo sequence, study medication will be placebo during the first phase (3 days) and during the second phase (3 days).
  For patients randomly assigned to the placebo/low-dose drug sequence, the patient will receive placebo for 3 days and then 10 mg/day CERC-501 for the following 3 days.
  For patients randomly assigned to the placebo/high-dose drug sequence, the patient will receive placebo for 3 days and then 20 mg/day CERC-501 for the following 3 days.
  Arms: Placebo/High-Dose Drug Arm; Placebo/Low-Dose Drug Arm; Placebo/Placebo Arm

SUMMARY:
This study is looking at the efficacy, rapidity, safety, and tolerability of two doses of oral CERC-501 for treating patients with treatment resistant depression who are taking an antidepressant that is not working for them.

DETAILED DESCRIPTION:
This study will involve 10 visits to the clinical site over approximately 1.5 months. There will be a screening visit (7-28 days may pass between the screening visit and the first treatment visit), a baseline/treatment visit (first day of study drug treatment), followed by 5 consecutive days of treatment visits. Follow-up visits will occur 6, 13, and 20 days after first receiving study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years old.
* Able to read, understand, and provide written, dated informed consent prior to screening.
* Diagnosed with Major Depressive Disorder (MDD), single or recurrent, and currently experiencing a Major Depressive Episode (MDE) of at least eight weeks in duration, prior to screening.
* Has a history of treatment resistance during the current MDE.
* Meet the threshold on the total MADRS score of greater than or equal to 20 at both screening and baseline visits, as confirmed by the remote centralized MGH CTNI rater between the screen visit and the baseline visit.
* In good general health
* For female participants, status of non-childbearing potential or use of an acceptable form of birth control
* Body mass index between 18-40 kg/m2
* Concurrent psychotherapy will be allowed if the type and frequency of the therapy has been stable for at least three months prior to screening and is expected to remain stable during participation in the study
* Concurrent benzodiazepine and hypnotic therapy will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

* Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study
* Female that is pregnant or breastfeeding
* Female with a positive pregnancy test at screening or baseline
* History during the current MDE of failure to achieve a satisfactory response to >3 treatment courses of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration during the current episode
* Total MADRS score of <20 at the screen or baseline visits, or as assessed by the remote, independent MGH CTNI rater and reported to the site
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence) with the exception of nicotine dependence, at screening or within six months prior to screening
* Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past 6 months or more)
* History of bipolar disorder, schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes
* History of eating disorders within five years of screening
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant at any time within 6 months prior to screening
* Subject is considered at significant risk for suicidal behavior during the course of their participation in the study
* Subject has had electroconvulsive therapy in the current episode of depression
* Has received vagus nerve stimulation (VNS) at any time prior to screening
* Dementia, delirium, amnestic, or any other cognitive disorder
* Has a clinically significant abnormality on the screening physical examination
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation
* Known history or current episode of: Uncontrolled hypertension, Recent myocardial infarction (within one year) or a history of more than one myocardial infarction, Syncopal event within the past year, Congestive heart failure, Angina pectoris, Systolic BP <85 or >160 mmHg or diastolic BP >95 mmHg or heart rate <50 or >105 beats per minute at screening or randomization, or QTcF greater than or equal to 450 msec at screening or randomization.
* Chronic lung disease
* Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder, epilepsy, mental retardation, or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system, or a history of significant head trauma within the past 2 years
* Presents with a history of Thyroid stimulating hormone outside of the normal limits and clinically significant as determined by the investigator
* Patients with diabetes mellitus fulfilling any of the following criteria:

  1. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.5% at screening
  2. Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus related illness in the past 12 weeks
  3. Not under physician care for diabetes mellitus
  4. Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.
  5. Any other clinically significant abnormal laboratory result (as determined after evaluation by study investigator and MGH CTNI medical monitor) at the time of the screening exam.
* History of hypothyroidism and has been on a stable dosage of thyroid replacement medication, or was surgically treated less than six months prior to screening
* History of hyperthyroidism which was treated (medically or surgically) less than six months prior to screening
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with the interpretation of study results
* History of positive screening urine test for drugs of abuse
* Patients with exclusionary laboratory values, or requiring treatment with exclusionary concomitant medications, including tricyclic antidepressants and monoamine oxidase inhibitors, or on two or more concomitant antidepressant therapies
* Patients currently taking a proton pump inhibitor (PPI)/histamine 2 (H2) blocker or with a history of chronic NSAID use
* Patients with a positive test for Helicobacter pylori (urea breath test)
* Patients with any of the following GI-related findings:

  1. Clinically evident GI complaints or GI disease at Screening or Visit 1
  2. Past history of gastric disease (including but not limited to peptic ulcer disease, gastritis (including atrophic gastritis), upper GI bleeding, any other GI precancerous conditions), and of any other clinically relevant GI disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2016-01-22 (Actual); Study Completion 2016-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital (Coordinating Center); Linda L Carpenter, MD, Principal Investigator — Brown University-Butler Hospital; John Zajecka, MD, Principal Investigator — Rush University; Mary F Morrison, MD, Principal Investigator — Temple University; Matthew Macaluso, DO, Principal Investigator — University of Kansas
Locations (4):
- United States (4):
  - Rush University, Chicago, Illinois
  - University of Kansas, Wichita, Kansas
  - Temple University, Philadelphia, Pennsylvania
  - Brown University-Butler Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 8 participants were randomized because the study terminated early due to slow enrollment.
Groups:
- Low Dose Drug-Drug Arm: Patients in this arm will receive CERC-501 10.0 mg/day for 3 days (in Phase 1) and for 3 subsequent days (in Phase 2)
  CERC-501: Low dose of CERC-501 will be 10 mg/day during the first phase (3 days) and during the second phase (3 days).
- High Dose Drug-Drug Arm: Patients in this arm will receive CERC-501 20.0 mg/day for 3 days (in Phase 1) and for 3 subsequent days (in Phase 2)
  CERC-501: High Dose of CERC-501 will be 20 mg/day during the first phase (3 days) and during the second phase (3 days).
- Placebo/Low-Dose Drug Arm: Patients in this arm will receive placebo for 3 days (in Phase 1) and CERC-501 10.0 mg/day for 3 days (in Phase 2)
  CERC-501: Low dose of CERC-501 will be 10 mg/day during the first phase (3 days) and during the second phase (3 days).
  For patients randomly assigned to the placebo/low-dose drug sequence, the patient will receive placebo for 3 days and then 10 mg/day CERC-501 for the following 3 days.
- Placebo/High-Dose Drug Arm: Patients in this arm will receive placebo for 3 days (in Phase 1) and CERC-501 20.0 mg/day for 3 days (in Phase 2)
  CERC-501: High Dose of CERC-501 will be 20 mg/day during the first phase (3 days) and during the second phase (3 days).
- Placebo/Placebo Arm: Patients in this arm will receive placebo for 3 days (in Phase 1) and for 3 subsequent days (in Phase 2)
  Placebo: For patients randomly assigned to the placebo/ placebo sequence, study medication will be placebo during the first phase (3 days) and during the second phase (3 days).
Period: Phase 1 (Days 0-2)
Arm/Group | Low Dose Drug-Drug Arm | High Dose Drug-Drug Arm | Placebo/Low-Dose Drug Arm | Placebo/High-Dose Drug Arm | Placebo/Placebo Arm
Started | 2 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Days 3-5)
Arm/Group | Low Dose Drug-Drug Arm | High Dose Drug-Drug Arm | Placebo/Low-Dose Drug Arm | Placebo/High-Dose Drug Arm | Placebo/Placebo Arm
Started | 2 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 8 participants were randomized because the study terminated early due to slow enrollment.
Groups:
- Placebo/Low-Dose Drug Arm: Patients in this arm will receive placebo for 3 days (in Phase 1) and CERC-501 10.0 mg/day for 3 days (in Phase 2)
  CERC-501: Low dose of CERC-501 will be 10 mg/day during the first phase (3 days) and during the second phase (3 days).
- Total: Total of all reporting groups
Arm/Group | Low Dose Drug-Drug Arm | High Dose Drug-Drug Arm | Placebo/Low-Dose Drug Arm | Placebo/High-Dose Drug Arm | Placebo/Placebo Arm | Total
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 8
Age, Continuous [Median (Full Range); unit: years] | 58.2 [52.1 to 64.4] | 58.3 [58.0 to 58.5] | 34.5 [34.5 to 34.5] | 36.3 [27.2 to 45.4] | 38.8 [38.8 to 38.8] | 48.8 [27.2 to 64.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 1 | 2 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 1 | 2 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 2 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 1 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression - 6 Items (HAM-D-6)
Description: This instrument is completed with a structured interview guide by the clinician based on his/her assessment of the patient's symptoms. This structured interview has been validated for use with time frames shorter than one week. Scale items are assessed based on symptoms within the past 24 hours. A higher score indicates more depression symptoms. Total scores range from 0 (normal) to 22 (severe).
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours after initiating treatment
Population: In the sequential parallel comparison design (SPCD) analyses through 72 hours, placebo non-responder data is included from phase 2 and is pooled with phase 1 data. All placebo participants from phase 1 were non-responders based on HAM-D-6 reduction and MADRS criteria.
Measure: Median (Full Range); unit: units on a scale
Groups:
- CERC-501: either dose (10 mg/day or 20 mg/day) of CERC-501; pooled patients from phase 1 and those on drug in phase 2 who were placebo non-responders from phase 1.
  Response is defined as a 50% or greater reduction from baseline to Day 3 on the Hamilton Rating Scale for Depression - 6 Items (HAM-D-6) total score and a Montgomery-Asberg Depression Rating Scale (MADRS) score of 16 or more at day 3.
- Placebo: Placebo therapy; pooled those on placebo in phase 1 with those on placebo in phase 2 who were placebo non-responders from phase 1.
  Response is defined as a 50% or greater reduction from baseline to Day 3 on the Hamilton Rating Scale for Depression - 6 Items (HAM-D-6) total score and a Montgomery-Asberg Depression Rating Scale (MADRS) score of 16 or more at day 3.
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale | -3 [-13.5 to 0] | 0 [-6 to 1.5]

2. Secondary Outcome: Change in Hamilton Rating Scale for Depression - 6 Items (HAM-D-6), Day 20
Description: as for outcome 1
Time Frame: Baseline and 20 days after initiating treatment
Population: The 20-day follow-up analyses only use drug-drug (either dose) and placebo-placebo arms. 2 participants were in low dose drug-drug arm, 2 participants were in high dose drug-drug arm, and 1 participant was in the placebo-placebo arm. One drug-drug pt missing day 20 data.
Measure: Median (Full Range); unit: units on a scale
Groups:
- CERC-501: either dose (10 mg/day or 20 mg/day) of CERC-501 in drug-drug arms
- Placebo: Placebo therapy in placebo-placebo arm
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 3 | 1
units on a scale | -3.5 [-5.5 to -0.5] | -3.5 [-3.5 to -3.5]

3. Secondary Outcome: Number of Participants With Response on Hamilton Rating Scale for Depression - 6 Items (HAM-D-6)
Description: Compare response rates at 72 hours for of patients treated with either dose (10 mg/day or 20 mg/day) of CERC-501 to those assigned to placebo therapy, using the Sequential Parallel Comparison Design (SPCD), with response defined as a 50% or greater reduction from baseline to Day 3 on the HAM-D-6 total score).
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
  The HAM-D-6 instrument is completed with a structured interview guide by the clinician based on his/her assessment of the patient's symptoms. This structured interview has been validated for use with time frames shorter than one week. Scale items are assessed based on symptoms within the past 24 hours. A higher score indicates more depression symptoms.
Time Frame: 72 hours after treatment initiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
Participants | 2 | 1

4. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The 10-item Montgomery-Asberg Depression Rating Scale (MADRS), which measures depression severity (in past 3 days), was completed by clinicians using an MGH structured interview. Each item is measured on a scale from 0 to 6, and the items are summed to find the total score. The total minimum score is 0 units on a scale and the total maximum score is 60 units on a scale, where higher scores indicate more severe depression.
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours and 20 days after initiating treatment
Population: In the sequential parallel comparison design (SPCD) analyses through 72 hours, placebo non-responder data is included from phase 2 and is pooled with phase 1 data. All placebo participants from phase 1 were non-responders based on HAM-D-6 and MADRS criteria. The 20-day follow-up analyses only use drug-drug (either dose) and placebo-placebo arms.
Measure: Median (Full Range); unit: units on a scale
Groups:
- CERC-501: For time frame through 72 hours: either dose (10 mg/day or 20 mg/day) of CERC-501; pooled patients from phase 1 and those on drug in phase 2 who were placebo non-responders from phase 1
  Response is defined as a 50% or greater reduction from baseline to Day 3 on the Hamilton Rating Scale for Depression - 6 Items (HAM-D-6) total score and a Montgomery-Asberg Depression Rating Scale (MADRS) score of 16 or more at day 3.
  For 20-day time frame: either dose drug-drug arms only
- Placebo: For time frame through 72 hours: Placebo therapy; pooled those on placebo in phase 1 with those on placebo in phase 2 who were placebo non-responders from phase 1.
  Response is defined as a 50% or greater reduction from baseline to Day 3 on the Hamilton Rating Scale for Depression - 6 Items (HAM-D-6) total score and a Montgomery-Asberg Depression Rating Scale (MADRS) score of 16 or more at day 3.
  For 20-day time frame: placebo-placebo arm only
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale
  72-hour change | -6.5 [-33 to 0] | -4.5 [-17 to 3]
  20-day change: number analyzed (Participants) | 3 | 1
  20-day change | -8 [-15.5 to -4.5] | -9 [-9 to -9]

5. Secondary Outcome: Change in Clinical Global Impression -Severity (CGI-S)
Description: The CGI-S scale was administered by clinicians to measure depressive severity (CGI-S). Each item is rated on a seven-point scale (1=normal to 7=among the most severe), so a higher total score indicates greater depressive severity. Severity is assessed based on the last 24 hours.
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours and 20 days after initiating treatment
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale
  72-hour change | -0.5 [-4 to 0] | 0 [-3 to 0.5]
  20-day change: number analyzed (Participants) | 3 | 1
  20-day change | -1 [-1.5 to 0] | -1 [-1 to -1]

6. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: The CGI-I scale was administered by clinicians to measure improvement in depressive severity (CGI-I). Each item is rated on a seven-point scale (1=very much improved to 7=very much worse), so a higher total score indicates less improvement in depressive severity. Improvement is assessed based on the last 24 hours.
Time Frame: 72 hours and 20 days after initiating treatment
Population: In the sequential parallel comparison design (SPCD) analyses through 72 hours, placebo non-responder data is included from phase 2 and is pooled with phase 1 data. All placebo participants from phase 1 were non-responders based on HAM-D-6 and MADRS criteria.The 20-day follow-up analyses only use drug-drug (either dose) and placebo-placebo arms.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale
  72 hours | 3 [1 to 4] | 4 [2 to 4]
  20 days: number analyzed (Participants) | 3 | 1
  20 days | 3 [3 to 4] | 4 [4 to 4]

7. Secondary Outcome: Change in Symptoms of Depression Questionnaire (SDQ)
Description: This validated self-rating instrument has 44 items on a scale of 1-6, measuring multiple depressive symptom domains. Each item is rated based on a subject's perception of what is normal for the individual (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). This scale is rated based on the past 24 hours. A total score is calculated by summing the 44 item scores, for a range of 0-264.
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours and 20 days after initiating treatment
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale
  72-hour change | -26 [-69.5 to 0] | -7.5 [-48 to 5]
  20-day change: number analyzed (Participants) | 3 | 1
  20-day change | -15.5 [-38.5 to -8.5] | -3.5 [-3.5 to -3.5]

8. Secondary Outcome: Change in Perceived Stress Scale (PSS)
Description: This is a 10-item, validated, self-rated measure of perceived stress, that is of the degree to which the subjects perceives things to be stressful and overwhelming. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. This scale is rated based on the past 24 hours.
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours and 20 days after treatment initiation
Population: In the sequential parallel comparison design (SPCD) analyses through 72 hrs, placebo non-responders are included from phase 2 and are pooled with phase 1. All placebo participants from phase 1 were non-responders based on HAM-D-6 and MADRS criteria. 2 pts missing 72-hr PSS values. The 20-day analyses only use drug-drug and placebo-placebo arms.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 6 | 4
units on a scale
  72-hour change | -3.5 [-13 to -1] | -1.25 [-2 to 2.5]
  20-day change: number analyzed (Participants) | 2 | 1
  20-day change | -7.25 [-12 to -2.5] | 0.5 [0.5 to 0.5]

9. Secondary Outcome: Change in Positive Affect Scale (PAS)
Description: This is a validated, self-rated measure of positive affect uses 5-point scales (1 = very slightly/not at all to 5 = extremely). Higher scores represent higher levels of positive affect. The scale is rated based on the past 24 hours. The total score is the sum of 10 items, for a range of 10-50.
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours and 20 days after initiating treatment
Population: In the sequential parallel comparison design (SPCD) analyses through 72 hrs, placebo non-responder data is included from phase 2 and is pooled with phase 1. All phase 1 placebo participants were non-responders based on HAM-D-6 and MADRS criteria.The 20-day analyses only use drug-drug (either dose) and placebo-placebo arms. 1 pt missing PAS data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale
  72-hour change | 8 [-5.5 to 19] | 17.5 [-25.5 to 31]
  20-day change: number analyzed (Participants) | 3 | 1
  20-day change | 11 [5 to 16.5] | 0 [0 to 0]

10. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Satisfaction With Participation in Social Roles and Discretionary Activities
Description: These are two well-validated 7-item self-rating scales that measure social health. A higher score represents higher satisfaction on each scale. The scales are rated based on the past 24 hours. Each item is rated 1-5 (1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much). Each 7-item subscale score is the sum of each of the 7 items and ranges from 7-35.
  To better estimate the baseline, we did not use simply the cross-sectional assessment at baseline, but we estimated the average during the screening period as the true baseline.
Time Frame: Baseline and 72 hours and 20 days after initiating treatment
Population: as for outcome 6
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale
  Social Roles 72-hour change | 2.5 [-4 to 11.5] | 1.5 [-4 to 11]
  Social Roles 20-day change: number analyzed (Participants) | 3 | 1
  Social Roles 20-day change | -1.5 [-3 to 7] | 3 [3 to 3]
  Discretionary Activities 72-hour change | 3 [0 to 16] | 1.5 [-2.5 to 6]
  Discretionary Activities 20-day change: number analyzed (Participants) | 3 | 1
  Discretionary Activities 20-day change | 4 [-1 to 7.5] | 5 [5 to 5]

11. Secondary Outcome: Change in the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS will be performed to assess suicidal ideation and behavior. It contains a 5-item rating scale for suicidal ideation and a 7-item rating scale for suicidal behavior. Higher total scores indicate higher severity. Each item is coded 1=yes, 0=no, so a total score of 0 on each scale means that a no response was entered for each of the 5 suicidal ideation and for each of the 7 suicidal behavior questions, i.e., 0=lowest severity score. Total suicidal ideation score ranges from 0 (least severe) to 5 (most severe). Total suicidal behavior score ranges from 0 (least severe) to 7 (most severe).
Time Frame: Baseline and 72 hours after initiating treatment
Population: In the sequential parallel comparison design (SPCD) analyses through 72 hours, placebo non-responder data is included from phase 2 and is pooled with phase 1 data. All placebo participants from phase 1 were non-responders based on HAM-D-6 reduction and MADRS criteria. 1 CERC-501 pt and 3 placebo pts are missing data on 72-hr change values.
Measure: Median (Full Range); unit: units on a scale
Groups:
- CERC-501: For time frame through 72 hours: either dose (10 mg/day or 20 mg/day) of CERC-501; pooled patients from phase 1 and those on drug in phase 2 who were placebo non-responders from phase 1
  Response is defined as a 50% or greater reduction from baseline to Day 3 on the Hamilton Rating Scale for Depression - 6 Items (HAM-D-6) total score and a Montgomery-Asberg Depression Rating Scale (MADRS) score of 16 or more at day 3.
- Placebo: For time frame through 72 hours: Placebo therapy; pooled those on placebo in phase 1 with those on placebo in phase 2 who were placebo non-responders from phase 1.
  Response is defined as a 50% or greater reduction from baseline to Day 3 on the Hamilton Rating Scale for Depression - 6 Items (HAM-D-6) total score and a Montgomery-Asberg Depression Rating Scale (MADRS) score of 16 or more at day 3.
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 6 | 2
units on a scale
  Suicidal Ideation | 0 [-2 to 0] | 0 [0 to 0]
  Suicidal Behavior | 0 [0 to 0] | 0 [0 to 0]

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal ECG
Description: Number of Participants with clinically significant abnormal electrocardiogram (ECG)
Time Frame: 72 hours after treatment initiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Labs
Description: Total number of participants with clinically significant abnormal labs
Time Frame: 72 hours after treatment initiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 7 | 5
Participants
  Total RBC | 1 | 1
  Hematocrit | 1 | 1
  Any lab | 1 | 1

ADVERSE EVENTS:
Groups:
- Low Dose Drug: Patients receive CERC-501 10.0 mg/day
- High Dose Drug: Patients receive CERC-501 20.0 mg/day
- Placebo: Patients receive placebo
Arm/Group | Low Dose Drug | High Dose Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Drug (N=3) | High Dose Drug (N=4) | Placebo (N=4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Central Nervous Systems Lesions (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disturbance (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Microscopic hematuria (grade 1) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Remembered dreams (unusual for subject) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Renal calculi (Grade 2) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
itching on thighs (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes